CLINICAL TRIAL: NCT00159380
Title: A Double Blind, Crossover Placebo-controlled Study to Evaluate the Effect of L-arginine and Aminoguanidine on Bronchial, Alveolar and Nasal NO and NO Metabolites
Brief Title: Nitric Oxide (NO) Donors and Inhibitors Study: Study to Evaluate L-Arginine and Aminoguanidine in Asthmatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2002AT033B
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — pimagedine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Healthy volunteers (Experimental): 8 non smokers non asthmatic
  Interventions: Drug: Placebos
- Asthma volunteers (Experimental): 8 asthmatic mild
  Interventions: Drug: Aminoguanidine

INTERVENTIONS:
Drug: Aminoguanidine — 500mg
  Other Names: Inhalation of aminoguanidine
  Arms: Asthma volunteers
Drug: Placebos — 2ml
  Other Names: Nebulase saline solution
  Arms: Healthy volunteers

SUMMARY:
The primary aim of this study is to investigate the effects of oral and inhaled administration of L-arginine and of inhaled aminoguanidine on bronchial and alveolar exhaled NO and NO metabolites in exhaled breath condensate, saliva and nasal lavage fluid in normal and asthmatic subjects.

DETAILED DESCRIPTION:
Nitric oxide (NO) is produced by a variety of cells within the respiratory tract, particularly airway epithelial cells, and its increased concentration in asthma is likely to derive from inducible NO synthase (iNOS) expressed in inflamed airways. To evaluate whether an increased bronchial flux of NO (ie, airway wall NO flux [Jno] in picoliters per second) produced in the large airways is due to an enzyme overexpression, we administered a relatively selective iNOS inhibitor, aminoguanidine, by nebulization in a double-blind, placebo-controlled manner in asthmatic and healthy subjects and also investigated whether the same concentration of inhibitor has any effect on NO produced in the peripheral lungs (ie, alveolar NO concentration [Calv] in parts per billion [ppb]) or on the diffusing capacity of NO (Dno) [in picoliters per second-1 per ppb-1) in the airways. Aminoguanidine administration resulted in a significant reduction in Jno compared with administration of the saline solution control in eight healthy subjects and in eight patients with asthma but caused no significant changes in Calv or in Dno in either group.

ELIGIBILITY:
Inclusion Criteria:

Healthy non-smokers (n=10):

* Nonatopic subjects (exhaled NO greater than or equal to 10 ppb; flow 50 ml/s)
* Normal spirometry
* Able to comprehend and grant a written informed consent

Asthmatic subjects (n=15):

* Forced expiratory volume in one second (FEV1) of no less than 70% of predicted (exhaled NO greater than or equal to 15 ppb; flow 50 ml/s)
* Clinically stable (steroid-naïve or taking no > 600 mcg/day of inhaled steroids)
* Able to comprehend and grant a written informed consent

Exclusion Criteria:

* Currently smoking
* Any lung disease other than asthma which may interfere with the study
* Treatment within the last 4 weeks with oral steroids
* Respiratory infection within 4 weeks prior to entry into the trial
* Females who are pregnant or lactating
* History of current or past drug or alcohol abuse

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Bronchial exhale nitric oxide | 6 hours
  Bronchial exhale nitric oxide (JNo) assessed by chemo luminescence
Peripheral exhaled nitric oxide | 6 hours
  Peripheral exhaled nitric oxide(CALV) assessed by chemo luminescence

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brindicci C, Ito K, Barnes PJ, Kharitonov SA. Effect of an inducible nitric oxide synthase inhibitor on differential flow-exhaled nitric oxide in asthmatic patients and healthy volunteers. Chest. 2007 Aug;132(2):581-8. doi: 10.1378/chest.06-3046. Epub 2007 Jun 5. PMID 17550932